CLINICAL TRIAL: NCT02356588
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of the Sublingual Sufentanil Tablet 30 mcg for the Treatment of Post-Operative Pain in Patients After Abdominal Surgery
Brief Title: A Trial Evaluating the Efficacy and Safety of the Sublingual Sufentanil Tablet 30 mcg for Post-Operative Pain After Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAP301
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sufentanil Tablet 30 mcg (Experimental): A stratified randomization will be applied in this study with sex as a stratification factor. Patients who meet all inclusion and none of the exclusion criteria at screening, and following surgery, will be randomly assigned at a 2:1 ratio to treatment with ST 30 mcg or PT within one of two groups (male or female) at each study center. Patients may receive a dose of study medication no more frequently than once per hour. The study may last up to 48 hours.
  Interventions: Drug: Sufentanil Tablet 30 mcg
- Placebo Tablet (Placebo Comparator): A stratified randomization will be applied in this study with sex as a stratification factor. Patients who meet all inclusion and none of the exclusion criteria at screening, and following surgery, will be randomly assigned at a 2:1 ratio to treatment with ST 30 mcg or PT within one of two groups (male or female) at each study center. Patients may receive a dose of study medication no more frequently than once per hour. The study may last up to 48 hours.
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Sufentanil Tablet 30 mcg
  Other Names: ST 30 mcg
  Arms: Sufentanil Tablet 30 mcg
Drug: Placebo Tablet
  Other Names: PT
  Arms: Placebo Tablet

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the sublingual Sufentanil Tablet (ST) 30 mcg to the sublingual Placebo Tablet (PT) for the short-term management of moderate-to-severe acute post-operative pain in patients after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria (additional criteria not specified here):

1. Patients who are scheduled to undergo one of the following procedures with general anesthesia or spinal anesthesia that does not include intrathecal opioids during the operation:

   * abdominoplasty
   * open tension-free inguinal hernioplasty (Lichenstein repair with mesh)
   * laparoscopic abdominal surgery
2. Patients classified as American Society of Anesthesiologists (ASA) class I - III (Appendix I).
3. Female patients of childbearing potential must be using an effective method of birth control at the time of screening visit
4. Patients who are expected to have moderate-to-severe post-operative pain for at least 24 hours.

Exclusion Criteria (additional criteria not specified here):

1. Patients who have taken an opioid for more than 30 consecutive days, at a daily dose of more than 15 mg of morphine (or equivalent), within the past 3 months prior to surgery
2. Patients who are currently taking monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 14 days of the first dose of study drug.
3. Patients with current sleep apnea that has been documented by a sleep laboratory study or are on home continuous positive airway pressure (CPAP).
4. Patients who previously have had abdominoplasty or have had an inguinal hernia repair on the same side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Palmer, M.D., PhD, Study Director — Talphera, Inc
Locations (4):
- United States (4):
  - Shoals Medical Trials, Inc, Sheffield, Alabama
  - Lotus Clinical Research, Pasadena, California
  - Victory Medical Center, Houston, Texas
  - Research Concepts, LLC, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Sufentanil Tablet 30 mcg: A stratified randomization will be applied in this study with sex as a stratification factor. Patients who meet all inclusion and none of the exclusion criteria at screening, and following surgery, will be randomly assigned at a 2:1 ratio to treatment with ST 30 mcg or PT within one of two groups (male or female) at each study center. Patients may receive a dose of study medication no more frequently than once per hour. The study may last up to 48 hours.
  Sufentanil Tablet 30 mcg
- Placebo Tablet: A stratified randomization will be applied in this study with sex as a stratification factor. Patients who meet all inclusion and none of the exclusion criteria at screening, and following surgery, will be randomly assigned at a 2:1 ratio to treatment with ST 30 mcg or PT within one of two groups (male or female) at each study center. Patients may receive a dose of study medication no more frequently than once per hour. The study may last up to 48 hours.
  Placebo Tablet
Period: Overall Study
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Started | 107 | 54
Completed | 102 | 41
Not Completed | 5 | 13
Not completed — Lack of Efficacy | 4 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet | Total
Number analyzed (Participants) | 107 | 54 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 106 | 53 | 159
  >=65 years | 1 | 1 | 2
Gender [Count of Participants; unit: Participants]
  Female | 73 | 36 | 109
  Male | 34 | 18 | 52

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 12-hour Study Period (SPID12).
Description: The primary outcome measure is the summed pain intensity difference to baseline over the 12-hour study period (SPID-12). A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and throughout the 12 hour study period. The SPID-12 is calculated by summing the difference between baseline pain score and pain score at each assessment time point.
  The observed SPID-12 scores ranged from -42.15 to 71.87 in the active group and -34.96 to 64.37 in the placebo group. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity.
Time Frame: 12 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
units on a scale | 25.84 (1.71) | 13.14 (2.35)

2. Secondary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 24-hour Study Period (SPID24).
Description: The primary outcome measure is the summed pain intensity difference to baseline over the 24-hour study period (SPID-24). A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and throughout the 24 hour study period. The SPID-24 is calculated by summing the difference between baseline pain score and pain score at each assessment time point. The observed SPID-24 scores ranged from -70.00 to 148.70 in the active group to -58.09 to 160.24 in the placebo group. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity.
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
units on a scale | 57.96 (3.45) | 37.28 (4.75)

3. Secondary Outcome: TOTPAR12
Description: Total pain relief over the 12 hours. The observed total pain relief scores ranged from 4.08 to 47.50 in the active group and 1.77 to 33.71 in the placebo group. A higher score indicates greater pain relief.
Time Frame: 12 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
units on a scale | 21.18 (0.87) | 15.36 (1.19)

4. Secondary Outcome: TOTPAR24
Description: Total pain relief over the 24 hour study period. The observed total pain relief scores ranged from 12.35 to 95.23 in the active group and 2.61 to 82.04 in the placebo group. A higher score indicates greater pain relief.
Time Frame: 24 Hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 102 | 41
units on a scale | 45.80 (1.81) | 35.45 (2.49)

5. Secondary Outcome: Time-weighted SPRID12
Description: Time-weighted summed pain relief intensity difference (SPRID) over the 12 hour study period. The observed SPRID scores ranged from -38.08 to 106.82 in the active group and -20.10 to 95.72 in the placebo group. A negative score indicates an increase in pain intensity and decrease in pain relief, while a higher score indicates a greater decrease in pain intensity and increase in pain relief.
Time Frame: 12 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 102 | 41
units on a scale | 47.03 (2.35) | 28.62 (3.24)

6. Secondary Outcome: Time-weighted SPRID24
Description: Time-weighted summed pain relief intensity difference (SPRID) over the 24 hour study period. The observed SPRID scores ranged from -49.67 to 222.04 in the active group and -24.97 to 237.54 in the placebo group. A negative score indicates an increase in pain intensity and decrease in pain relief, while a higher score indicates a greater decrease in pain intensity and increase in pain relief.
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 102 | 41
units on a scale | 103.88 (4.81) | 73.05 (6.62)

7. Secondary Outcome: Patient Global Assessment
Description: Proportion of patients who responded good or excellent to the global assessment of method of pain control at 24 hours
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 102 | 41
Percentage of patients | 80.4 [72.85 to 91.37] | 51.9 [38.52 to 65.18]

8. Secondary Outcome: Healthcare Professional Global Assessment
Description: Proportion of Health Care Professionals who responded good or excellent to the global assessment of method of pain control at 24 hours
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: Percentage of HCPs
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
Percentage of HCPs | 80.4 [72.85 to 87.90] | 53.7 [40.40 to 67.00]

9. Secondary Outcome: Summed Pain Intensity Difference
Description: The SPID-1 is calculated by summing the difference to baseline between baseline pain score and the pain score at each assessment time point through 1 hour.
  The observed SPID scores ranged from -2.00 to 5.25 in the active group to -4.90 to 3.00 in the placebo group. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity.
Time Frame: 1 hour
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
units on a scale | 1.09 (0.15) | -0.37 (0.21)

10. Secondary Outcome: Analysis of Total Number of Doses Used During the 12-Hour Study Period in the ITT Population
Time Frame: Cumulative through 12 hours
Measure: Mean (Standard Deviation); unit: mean number of tablets taken
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
mean number of tablets taken | 4.4 (2.0) | 4.7 (2.3)

11. Secondary Outcome: Analysis of Total Number of Doses Used During the 24-Hour Study Period in the ITT Population
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mean number of tablets taken
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
mean number of tablets taken | 7.09 (3.60) | 6.40 (3.80)

12. Secondary Outcome: Summary of Number of Rescue Morphine Doses Used by Study Period in the ITT Population
Time Frame: Cumulative through 6 hours
Measure: Mean (Standard Deviation); unit: mean number of doses used
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 57
mean number of doses used | 0.3 (0.7) | 1.1 (1.1)

13. Secondary Outcome: Summary of Number of Rescue Morphine Doses Used by Study Period in the ITT Population
Time Frame: Cumulative through 12 hours
Measure: Mean (Standard Deviation); unit: mean number of doses used
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
mean number of doses used | 0.4 (1.0) | 1.6 (1.8)

14. Secondary Outcome: Summary of Number of Rescue Morphine Doses Used by Study Period in the ITT Population
Time Frame: Cumulative through 24 hours
Measure: Mean (Standard Deviation); unit: mean number of doses used
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Number analyzed (Participants) | 107 | 54
mean number of doses used | 0.5 (1.4) | 2.1 (2.9)

ADVERSE EVENTS:
Time Frame: Non serious adverse events reported 12 hours after the first dose of study drug was given were recorded; SAEs reported within 30 days of last dose of study drug were recorded.
Arm/Group | Sufentanil Tablet 30 mcg | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 0/107 | 2/54
Other Adverse Events (participants affected / at risk) | 49/107 | 21/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil Tablet 30 mcg (N=107) | Placebo Tablet (N=54)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil Tablet 30 mcg (N=107) | Placebo Tablet (N=54)
Nausea (Gastrointestinal disorders) | 31 | 12 — The AEs listed in this table are those recorded as possibly or probably related to study drug
Headache (Nervous system disorders) | 13 | 6
Dizziness (Nervous system disorders) | 6 | 2
Hypotension (Cardiac disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 6 | 1
Nausea, Procedural (Gastrointestinal disorders) | 3 | 2
Somnolence (Nervous system disorders) | 3 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other